CLINICAL TRIAL: NCT06350812
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Multiple Dose Escalating Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PB-119 Injection in Chinese Obese Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PB-119 Injection in Chinese Obese Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PegBio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PB119110
Record Dates: First submitted 2024-03-18; First posted 2024-04-05 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PB-119 (Experimental): PB-119 administered on the first day of week 1-20 according to the dose-escalation design
  Interventions: Drug: PB-119
- Placebo (Placebo Comparator): Matched placebo administered on the first day of week 1-20 according to the dose-escalation design
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PB-119 — Administered subcutaneously once a week
  Arms: PB-119
Drug: Placebo — Administered subcutaneously once a week
  Arms: Placebo

SUMMARY:
The trial is conducted in a single-center, randomized, double-blind, placebocontrolled, dose-increasing design. To evaluate the safety, tolerability, pharmacokinetics(PK) characteristics, efficacy and immunogenicity of PB-119 injection in Chinese obese subjects.

DETAILED DESCRIPTION:
The trial is conducted in a single-center, randomized, double-blind, placebocontrolled, dose-increasing design. To evaluate the safety, tolerability, PK characteristics, efficacy and immunogenicity of PB-119 injection in Chinese obese subjects. The study consists of 1-2 cohort . 32 patients are planned to be included in each cohort (24 patients receive study drug，8 patients receive placebo) Subjects will receive treatment for 20 weeks after screening and complete 4 weeks of safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male or female subjects aged 18-60 years (both inclusive).
2. Body weight ≥70 kg(male) or 60 kg(female), and body mass index (BMI)

   ≥30.0 kg/m2 at screening.
3. Weight change <5% in the past 3 months before screening.

Exclusion Criteria:

1. Fasting Plasma Glucose（FPG） ≥7.0mmol/L or glycosylated hemoglobin (HbA1c) ≥6.5% or diagnosed diabetes
2. FPG <3.9 mmol/L at screening and/or a history of hypoglycemia.
3. History of Cushing's syndrome, polycystic ovaries, or other hereditary endocrine disorders, or obesity caused by secondary factors such as cortisol hormones.
4. Abnormal Thyroid-Stimulating hormone(TSH), Serum Free Triiodothyronine（FT3）, Serum Free Thyroxine（FT4） or diagnosed thyroid dysfunction
5. History of multiple endocrine neoplasia syndrome type 2 (MEN-2) , medullary thyroid carcinoma (MTC) or Category 4 and above thyroid nodules by Thyroid ultrasound Chinese Ultrasound Thyroid Imaging Reporting and Data System （C-TIRADS）
6. Diagnosed cardiovascular and cerebrovascular diseases with obvious clinical significance within 6 months before screening
7. Systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg at screening or randomization.
8. Time history from the starting point of P-wave to the starting point of QRS wave（PR intervals ）> 210 msec and/or QRS complex（QRS） > 120 msec and/or Corrected QT Interval（QTcF） > 450 msec at screening or randomization.
9. Serum amylase or lipase > 3× upper limit of normal (ULN) at screening or before randomization, or previously diagnosed acute/chronic pancreatitis.
10. Low density lipoprotein cholesterol(LDL-C) ≥4.40 mmol/L or triglyceride (TG) ≥5.65 mmol/L.
11. Use of any approved or unapproved drugs or products that have an effect on body weight within 3 months prior to screening
12. History of bariatric surgery for weight loss before screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From the first dosing (Day 1 ) of study drug until completion of the post treatment follow-up visit (24 week)

SECONDARY OUTCOMES:
Pharmacokinetic profile | From the first dose (Day 1 ) of study drug until 20 week
  Cmax
Pharmacokinetic profile | From the first dose (Day 1 ) of study drug until 20 week
  Tmax
Pharmacokinetic profile | From the first dose (Day 1 ) of study drug until 20 week
  area under the curve0(AUC0)-tau
Pharmacokinetic profile | From the first dose (Day 1 ) of study drug until 20 week
  AUC0-last
Effectiveness index | week 20
  Change in body weight from baseline
Effectiveness index | week 20
  Proportion of participants with ≥5% weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Yang, Ph D, Principal Investigator — The Third Xiangya Hospital of Central South University; Ping Jin, Ph D, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third XIANGYA Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No